Effect of lymphedema prevention program based on theory of Knowledge-attitude-practice on postoperative breast cancer patients: a randomized clinical trial

Research Proposal

(Version date: May 4, 2021)

Unique Protocol ID:19900601

## **Data Analysis**

SPSS21.0 software was used, a two-sided test was set, and  $\,^\alpha\,$  was set at 0.05.The normality of measurement data was expressed as mean  $\,^\pm\,$  standard deviation ( $\,^\pm\,$ s), and two independent sample t-test was used. When not normal, the median and interquartile range [M(Q)] were expressed using the Mann-Whitney U test. Enumeration data were expressed as frequency and constituent ratio using 2 test. Mann-whitney U test was used for grade data.

Table 1 Socio-demographic and clinical characteristics at baseline, by group allocation

| | | Total | Intervention Group | Control Group | |
|---|---|---|---|---|---|
| Characteristics | | (n=97) | ( <i>n</i> =47) | ( <i>n</i> =50) | $t/Z/X^2$ P |
| Age (X±SD) | | 50.51±9.78 | 50.15±11.01 | 50.84±8.56 | -0.344 0.732° |
| BMI (X±SD) | | 23.50±2.81 | 23.32±2.78 | 23.67±2.86 | -0.620 0.536 |
| Marital status (%) | Married | 91 (93.8) | 44 (93.6) | 47 (94.0) | -1.597 0.899° |
| , | Never married | 1 (1.0) | 1 (2.1) | 0 (0.0) | |
| | Divorced | 3 (3.1) | 1 (2.1) | 2 (4.0) | |
| | Widowed | 2 (2.1) | 1 (2.1) | 1 (2.0) | |
| Education level (%) | Junior high school or below | 42 (43.3) | 21 (44.7) | 21 (42.0) | 0.282 0.778 <sup>t</sup> |
| | High school or<br>technical<br>school | 25 (25.8) | 12 (25.5) | 13 (26.0) | |
| | College or above | 30 (30.9) | 14 (29.8) | 16 (32.0) | |
| Occupation (%) | Enterprise personnel | 18 (18.6) | 10 (21.3) | 8 (16.0) | -2.156 0.827° |
| | Peasantry | 29 (29.9) | 14 (29.8) | 15 (30.0) | |
| | Merchant | 15 (15.5) | 8 (17.0) | 7 (14.0) | |
| | Technicist | 13 (13.4) | 4 (8.5) | 9 (18.0) | |
| | Unemployed | 12 (12.4) | 6 (12.8) | 6 (12.0) | |
| | Others | 10 (10.3) | 5 (10.6) | 5 (10.0) | |
| Monthly incom<br>(RMB) (%) | e<br><1500 | 16 (16.5) | 8 (17.0) | 8 (16.0) | 0.316 0.752 <sup>b</sup> |
| | 1500-3000 | 35 (36.1) | 17 (36.2) | 18 (36.0) | |
| | 3001-5000 | 25 (25.8) | 13 (27.7) | 12 (24.0) | |
| | >5000 | 21 (21.6) | 9 (19.1) | 12 (24.0) | |
| Affected extremit | ty<br>Left | 45 (46.4) | 19 (40.4) | 26 (52.0) | -1.305 0.253° |
| | Right | 52 (53.6) | 28 (59.6) | 24 (48.0) | |
| Disease stage (%) | I | 38 (39.2) | 23 (48.9) | 15 (30.0) | 1.630 0.103 <sup>t</sup> |
| | II | 43 (44.3) | 17 (36.2) | 26 (52.0) | |

| | III | 16 (16.5) | 7 (14.9) | 9 (18.0) | |
|---|---|---|---|---|---|
| Operation type (%) | Mastectomy | 75 (77.3) | 36 (76.6) | 39 (78.0) | -0.380 0.931 <sup>c</sup> |
| | Conserving surgery | 17 (17.5) | 8 (17.0) | 9 (18.0) | |
| | Mastectomy and rebuild | 5 (5.2) | 3 (6.4) | 2 (4.0) | |
| Number of axillar lymph node extracted [M(Q)] | • | 5.00 (3.00, 19.00) | 7.00 (3.00, 21.00) | 5.00 (3.00, 17.30) | 0.962 0.336 <sup>b</sup> |
| Time of drainag<br>tube extraction (day<br>[M(Q)] | | 9.00 (7.00, 12.50) | 8.00 (7.00, 14.00) | 10.00 (7.00, 12.00) | 0.125 0.901 <sup>b</sup> |

Note: a Independent sample test.

<sup>b</sup>Mann-Whitney U test.

<sup>c</sup>Chi-square test.

Table 2 Comparison of upper limb lymphedema incidence between two groups after intervention

| - | Post-test1 (T1) | | | | Post-test2 (T2) | | | |
|---|---|---|---|---|---|---|---|---|
| Lymphedema | Intervention | Control | $\chi_2$ | Р | Intervention | Control | χ2 | Р |
| | (n=47) | (n=50) | | | (n=47) | (n=50) | | |
| None (%) | 46 (97.9) | 48 (96.0) | | 1.000 | 45 (95.7) | 46 (92.0) | | |
| Total (%) | 1 (2.1) | 2 (4.0) | 0.000 | | 2 (4.3) | 4 (8.0) | 0.118 | 0.731 |

 $<sup>\</sup>chi^2$ =Chi-square test.

Table 3 Comparison of the severity of upper limb lymphedema between two groups after intervention

| _ | Post-test1 (T1) | | _ | Post-test2 (T2) | | | _ | |
|---|---|---|---|---|---|---|---|---|
| Lymphedema | Intervention | Control | Z | Ρ | Intervention | Control | Z | Р |
| | (n=47) | ( <i>n</i> =50) | | | (n=47) | ( <i>n</i> =50) | | |
| None (%) | 46 (97.9) | 48 (96.0) | | | 45 (95.7) | 46 (92.0) | | |
| Mild (%) | 1 (2.1) | 2 (4.0) | 0.530 | 0.596 | 2 (4.3) | 3 (6.0) | 0.752 | 0.452 |
| Moderate | 0 (0.0) | 0 (0.0) | | | 0 (0.0) | 1 (2.0) | | |

| Severe (%) | 0 (0.0) | 0 (0.0) | 0 (0.0) | 0 (0.0) |
|--------------|---------|---------|---------|---------|
| 30 00 0 (70) | 0 (0.0) | 0 (0.0) | 0 (0.0) | 0 (0.0) |

z=Mann-Whitney U test.

Table 4 Comparison of handgrip strength between two groups after intervention

| Group | Pre-test (T0) | Post-test1 (T1) | Post-test2 (T2) | Group | Time | Group × time | D2* |
|---|---|---|---|---|---|---|---|
| | X±SD | X±SD | X±SD | F (P) | F (P) | F (P) | - ηP <sup>2</sup> * |
| Intervention | 22.02±5.78 | 18.04±5.77 | 21.48±5.65 | 1.975 | 243.426 | 27.665 | 0.271 |
| Control | 22.16±5.25 | 16.18±4.22 | 19.21±4.30 | (0.163) | (<0.001) | (<0.001) | 0.371 |
| t | 0.122 | -2.172 | -2.232 | | | | |
| P | 0.903 | 0.032 | 0.028 | | | | |

t=Independent sample test.

Table 5 Comparison of ROM between two groups after intervention

| Croup | Pre-test (T0) | Post-test1 (T1) | Post-test2 (T2) | Group | Time | Group × time | ~ D2* |
|---|---|---|---|---|---|---|---|
| Group | X±SD | X±SD | X±SD | F (P) | F (P) | F (P) | · ηP <sup>2</sup> * |
| Flexion | | | | | | | |
| Intervention | 21.26±5.49 | 119.87±20.49 | 146.74±16.10 | 10.646 | 2332.200 | 3.289 | 0.065 |
| Control | 19.21±4.30 | 107.54±24.03 | 136.74±18.93 | (0.002) | (<0.001) | (0.042) | 0.065 |
| t | -2.058 | -2.712 | -2.952 | | | | |
| P | 0.042 | 0.008 | 0.004 | | | | |
| Extension | | | | | | | |
| Intervention | 60.21±7.79 | 51.53±10.23 | 59.96±9.71 | 3.941 | 70.293 | 1.256 | 0.026 |
| Control | 58.12±8.31 | 46.74±10.35 | 53.80±8.87 | (0.050) | (<0.001) | (0.290) | 0.026 |
| t | -1.293 | -2.292 | -0.674 | | | | |
| P | 0.199 | 0.024 | 0.097 | | | | |
| Abduction | | | | | | | |
| Intervention | 160.34±11.99 | 120.60±20.51 | 147.51±16.99 | 9.893 | 190.291 | 7.038 | 0.130 |

<sup>\*=</sup>The effect size of the interact (group  $\times$  time) effect.

| Control | 160.20±11.72 | 107.4±25.91 | 132.26±23.07 | (0.002) | (<0.001) | (0.001) | |
|---|---|---|---|---|---|---|---|
| t | -0.058 | -2.770 | -3.722 | | | | |
| P | 0.954 | 0.007 | <0.001 | | | | |
| Adduction | 0.50 . | 0.007 | 10.001 | | | | |
| Intervention | 50.43±8.52 | 45.00±8.19 | 48.87±8.24 | 0.054 | 40.095 | 0.472 | 0.005 |
| Control | 49.90±6.43 | 45.30±7.60 | 48.12±6.69 | (0.817) | (<0.001) | (0.625) | |
| t | -0.341 | 0.187 | -0.495 | | | | |
| Р | 0.734 | 0.852 | 0.622 | | | | |
| Internal rotation | n | | | | | | |
| Intervention | 53.83±7.39 | 51.15±8.94 | 53.47±7.33 | 0.388 | 11.885 | 2.833 | 0.057 |
| Control | 53.76±7.06 | 50.50±7.09 | 51.66±6.15 | (0.535) | (<0.001) | (0.064) | 0.057 |
| t | -0.048 | -0.397 | 1.319 | | | | |
| Р | 0.962 | 0.692 | 0.190 | | | | |
| External rotatio | n | | | | | | |
| Intervention | 64.19±10.65 | 55.79±9.73 | 62.21±10.39 | 1.292 | 60.940 | 2.302 | 0.047 |
| Control | 62.86±11.05 | 53.60±10.54 | 58.96±10.36 | (0.259) | (<0.001) | (1.106) | 0.047 |
| t | -0.604 | -1.060 | -1.534 | | | | |
| P | 0.548 | 0.292 | 0.126 | | | | |

t=Independent sample test.

Table 6 Comparison of DASH scores between two groups after intervention

| Group | Pre-test (T0) | Post-test1 (T1) | Post-test1 (T2) | Group | Time | Group × time | D2* |
|---|---|---|---|---|---|---|---|
| | X±SD | X±SD | X±SD | F (P) | F (P) | F (P) | - ηP <sup>2</sup> * |
| Intervention | 3.00±4.40 | 29.84±12.47 | 11.65±6.71 | 18.978 | 296.757 | 11.685 | 0.100 |
| Control | 3.23±3.35 | 38.00±16.19 | 18.23±6.65 | (<0.001) | (<0.001) | (<0.001) | 0.199 |
| t | 0.290 | 2.770 | 4.845 | | | | |
| P | 0.773 | 0.007 | <0.001 | | | | |

 $t \hbox{=} Independent \ sample \ test.$ 

<sup>\*=</sup>The effect size of the interact (group  $\times$  time) effect.

<sup>\*=</sup>The effect size of the interact (group  $\times$  time) effect.

Table 7 Comparison of FACT-B scores between two groups after intervention

| Communication | Pre-test (T0) | Post-test1 (T1) | Post-test2 (T2) | Group | Time | Group × time | D?* |
|---|---|---|---|---|---|---|---|
| Group | X±SD | X±SD | X±SD | F (P) | F (P) | F (P) | - ηP <sup>2</sup> * |
| Physical well-be | eing | | | | | | |
| Intervention | 22.81±3.25 | 18.04±3.31 | 21.19±3.49 | 2.789 | 46.483 | 0.244 (0.000) | 0.005 |
| Control | 22.50±4.49 | 17.36±3.37 | 20.12±4.06 | (0.098) | (<0.001) | 0.214 (0.808) | 0.005 |
| t | -0.390 | -1.006 | -1.390 | | | | |
| P | 0.698 | 0.317 | 0.168 | | | | |
| Social/family w | ell-being | | | | | | |
| Intervention | 19.57±3.90 | 18.34±4.86 | 19.58±1.87 | 7.639 | 5.483 | 1.670 (0.194) | 0.034 |
| Control | 19.28±4.27 | 16.33±4.87 | 17.71±2.71 | (0.007) | (0.006) | 1.670 (0.194) | 0.034 |
| t | -0.364 | -2.038 | -3.983 | | | | |
| P | 0.730 | 0.044 | <0.001 | | | | |
| Emotional well- | -being | | | | | | |
| Intervention | 14.19±3.52 | 17.26±3.67 | 18.13±2.59 | 17.418 | 25.944 | 1.463 (0.234) | 0.015 |
| Control | 13.60±2.39 | 15.42±2.81 | 16.06±3.79 | (<0.001) | (<0.001) | | 0.013 |
| t | -0.963 | -2.749 | -3.151 | | | | |
| Р | 0.339 | 0.077 | 0.002 | | | | |
| Functional well | -being | | | | | | |
| Intervention | 17.23±4.86 | 16.60±5.12 | 18.34±2.10 | 7.328 | 6.316 | 1.516 (0.225) | 0.031 |
| Control | 17.28±5.36 | 14.44±3.79 | 16.38±3.88 | (800.0) | (0.003) | 1.510 (0.225) | 0.031 |
| t | 0.044 | -2.344 | -3.123 | | | | |
| Р | 0.965 | 0.021 | 0.003 | | | | |
| Breast cancer s | ession | | | | | | |
| Intervention | 29.02±2.19 | 22.81±3.34 | 25.53±3.16 | 10.276 | 174.609 | 7.649 (0.001) | 0.137 |
| Control | 29.34±2.80 | 21.42±3.73 | 22.82±4.38 | (0.002) | (<0.001) | 7.045 (0.001) | 0.137 |
| t | 0.622 | -1.928 | -3.476 | | | | |
| P | 0.535 | 0.057 | 0.001 | | | | |
| Total | | | | | | | |

| Intervention | 102.83±11.25 | 93.05±11.15 | 102.77±8.66 | 19.425 | 39.240 | 4 606 (0.010) | 0.047 |
|---|---|---|---|---|---|---|---|
| Control | 102.00±12.98 | 84.97±10.03 | 93.09±12.22 | (<0.001) | (<0.001) | 4.696 (0.010) | 0.047 |
| t | -0.333 | -3.754 | -4.525 | | | | |
| Р | 0.740 | <0.001 | <0.001 | | | | |

t=Independent sample test.

<sup>\*=</sup>The effect size of the interact (group  $\times$  time) effect.